CLINICAL TRIAL: NCT07406854
Title: A Phase 3, Multicenter, Randomized, Double-Masked, Sham-Controlled Clinical Trial to Evaluate the Safety and Efficacy of Gene Therapy for Leber's Hereditary Optic Neuropathy (LHON) Associated With ND4 Mutation
Brief Title: A Phase 3, Multicenter, Randomized, Double-Masked, Sham-Controlled Clinical Trial for Leber's Hereditary Optic Neuropathy (LHON) Associated With ND4 Mutation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wuhan Neurophth Biotechnology Limited Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFS-01-201
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Leber Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-Masked, Sham-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: NR082 injection (Experimental): 4.5E9 viral genomes (vg) , 0.05 mL eye/dose , bilaterally
  Interventions: Genetic: rAAV2-ND4
- Sham Comparator: sham-injection (Sham Comparator): Sham intravitreal injection （bilateral）will be performed by applying pressure to the eye at the location of a typical intravitreal injection procedure using the blunt end of a syringe without a needle.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Genetic: rAAV2-ND4 — a single bilateral intravitreal (IVT) injection of NR082
  Arms: Experimental: NR082 injection
Other: Sham (No Treatment) — sham-injection
  Arms: Sham Comparator: sham-injection

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of NR082 in the treatment of LHON caused by mitochondrial ND4 gene mutation. This study will enroll subjects aged ≥ 12 years old and ≤ 75 years old to receive a single bilateral intravitreal (IVT) injection of NR082 to evaluate safety and efficacy. The clinical manifestations of all subjects are to be reduced visual acuity caused by LHON associated with ND4 mutation, with laboratory test showing G11778A mutation and reduced visual acuity lasted for >6 months and <10 years.

DETAILED DESCRIPTION:
Safety run-in phase:

The safety run-in phase will enroll 6 evaluable subjects aged ≥ 12 years and ≤ 75 years , namely 4.5 x 109 vg, 0.05 mL eye/dose（bilaterally） and monitor the safety for at least 6 weeks. If there is no new safety concern evaluated by the SRC, the randomized, double-blind, sham-injection control study can be initiated.

Second Stage: randomized, double-blind, sham-injection control study:

The randomized, double-blind, sham-injection control study is to verify the efficacy and safety of NR082 in LHON caused by mitochondrial gene ND4 mutation . This part is divided into the NR082 treatment group and the control group (sham-injection group).

ELIGIBILITY:
Inclusion Criteria:

* Age at the time of signing the informed consent form: the age of the subjects must be ≥ 12 years old and ≤ 75 years old
* The clinical manifestation of all subjects is reduced visual acuity caused by LHON associated with ND4 mutation, while the reduced visual acuity lasted for > 6 months and < 10 years
* The clinical manifestation caused by LHON is vision loss, with a visual acuity of ≥ 0.5 LogMAR and ≤1.68 in BCVA in both eye The genotype test result is that there is G11778A mutation in ND4 gene, and there are no other primary LHON-associated mutations in the mitochondrial DNA (mtDNA) (ND1[G3460A] or ND6[T14484C]) (confirmed by a CLIA-certified international laboratory) Pupils can be adequately dilated for a comprehensive eye examination and visual acuity test

Exclusion Criteria:

* Any known allergy and/or hypersensitivity to the study drug or its constituents Contraindication to IVT injection in any eye
* IVT drug delivery to any eye within 30 days prior to the screening visit History of vitrectomy in either eye
* Narrow anterior chamber angle in any eye contra-indicating pupillary dilation
* Presence of disorders or diseases of the eye or adnexa, excluding LHON, which may interfere with visual or ocular assessments, including optical coherence tomography during the study
* Presence of known/documented mutations, other than the LHON-related mutation, which are known to cause pathology of the optic nerve, retina or afferent visual system
* Presence of systemic or ocular/vision diseases, disorders or pathologies, other than LHON, known to cause or be associated with vision loss, or whose associated treatment(s) or therapy(ies) is/are known to cause or be associated with vision loss
* Presence of optic neuropathy from any cause other than LHON
* Presence of illness or disease that, in the opinion of the investigator, include symptoms and/or the associated treatments that can alter visual function, for instance cancers or pathology of the CNS, including multiple sclerosis (diagnosis of multiple sclerosis must be based on the 2010 Revisions to the McDonald Criteria) (Polman et al., 2011), and/or diseases or conditions that affect the safety of subjects participating in the study
* History of recurrent uveitis (idiopathic or immune-related) or active ocular inflammation
* Participated in another clinical study and receive IP within 90 days prior to the screening visit

  a) Exceptions: Subjects who have completed the clinical study of idebenone as IP within 90 days prior to the screening visit, and has completely discontinued idebenone at least 7 days prior to dosing are still eligible to participate in the study.
* Any eye has previously received ocular gene therapy
* Subjects who refused to stop using idebenone
* Have undergone ocular surgery of clinical relevance (per investigator's assessment) within 90 days prior to the screening visit
* Female subjects who are breastfeeding or plan to breastfeed within the first 6 months after the administration of NR082 Injection
* History of drug or alcohol abuse (including heavy smoking, i.e. > 20 cigarettes per day or > 20 pack-years [equivalent to one pack a day for 20 years or 2 packs a day for 10 years])
* Subjects with positive human immunodeficiency virus (HIV), syphilis and HCV antibodies are excluded; subjects who have clinically significant active infection requiring treatment as shown by hepatitis B test (defined as positive hepatitis B core antibody [HBcAb] or hepatitis B surface antigen [HBsAg], hepatitis B virus deoxyribonucleic acid (HBV-DNA) >1,000 copies /mL or >lower limit of quantitative detection with the local laboratory method) will be excluded
* Unable to tolerate or unable or unwilling to comply with all the protocol requirements
* Any other exclusions determined by the investigator

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of NR082 in study eye | 52 weeks
  Proportion of ≥ 0.3 LogMAR from baseline in BCVA in the study eye in the NR082 treatment and the sham-injection at Week 52 after treatment

SECONDARY OUTCOMES:
Efficacy of NR082 in study eye and non-study eye | 52 weeks
  Mean change from baseline in BCVA;
Mean change from baseline in visual field, contrast sensitivity | 52 weeks
  Efficacy of NR082 in study eye and non-study eye
Safety and tolerability of NR082 | 52 weeks
  Incidence rates of AEs, SAEs within 52 weeks after injection of NR082

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No